CLINICAL TRIAL: NCT01252082
Title: Evaluation of Effect of Nonsurgical Periodontal Therapy on Metabolic Control in Patients With Type II Diabetes
Brief Title: Non-surgical Periodontal Therapy Effects Metabolic Control in Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Moeintaghavi, associate professor of periodontics, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 86067
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Metabolic Control
Keywords: metabolic control; fasting plasma glucose; glycated hemoglobin
MeSH Terms: interventions — Tooth Exfoliation; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scalig and Rootplaning (Active Comparator): patients will receive scaling and root planing therapy
  Interventions: Procedure: Scaling and Rootplaning
- control (No Intervention): patients in control group will not receive periodontal treatment in the time period of the study

INTERVENTIONS:
Procedure: Scaling and Rootplaning — All patients in the test group receive scaling and rootplaning under local anesthesia
  Other Names: test group; control group
  Arms: Scalig and Rootplaning

SUMMARY:
The purpose of this study is to determine whether nonsurgical periodontal therapy is effective in the metabolic control of patients with type II Diabetes mellitus.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (DM2), the most common type of diabetes, is characterized by hyperglycemia, hyperlipidemia, and associated complications. The classic major complications of diabetes are microangiopathy, nephropathy, neuropathy, macrovascular disease, delayed wound healing, and periodontitis. There is an interacting, complex relationship between diabetes and periodontitis.Many studies have shown a greater incidence and a greater severity of periodontitis in diabetic patients.Meanwhile, a number of studies have suggested that periodontitis may actually be a risk factor for diabetic complications as well. This study is performed to investigate the effects of non-surgical periodontal therapy on metabolic control in DM2 patients.

ELIGIBILITY:
Inclusion Criteria:

(1) mild to moderate periodontitis according to the criteria of the American Academy of Periodontology (32); (2) diagnosis of DM2 with glycated hemoglobin (HbA1c) values over 7%; (3) no major diabetic complications; (4) blood sugar controlled with glybenclamide and metformin, without insulin administration; and (5) no systemic antibiotic administration or periodontal treatment within the last 6 months.

Exclusion Criteria:

(1) presence of systemic diseases other than DM2 that may influence the course of periodontal disease; (2) intake of immunosuppressive drugs, steroids, hydantoin, or non-steroidal anti-inflammatory drugs; (3) tobacco use; (4) pregnancy or intention to become pregnant during the study period; (5) fixed orthodontic appliances; and (5) refusal or inability to give informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Metabolic control | 3 months after treatment
  fasting plasma glucose (FPG), HbA1c, TG, TC, high density lipoprotein cholesterol (HDL), and LDL are measured at baseline and 3 months after treatment.

SECONDARY OUTCOMES:
periodontal improvement after scaling and rootplaning | 3 months after treatment
  Periodontal parameters (Plaque index, Gingival index, Clinical Attachment level and Probing depth)are Measured at baseline and 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moeintaghavi, DDS.,Ms., Study Chair — Associate professor,Mashhad Dental School, Mashhad University of Medical Sciences
Locations (1):
- Mashhad Dental School, Mashhad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Result] Moeintaghavi A, Arab HR, Bozorgnia Y, Kianoush K, Alizadeh M. Non-surgical periodontal therapy affects metabolic control in diabetics: a randomized controlled clinical trial. Aust Dent J. 2012 Mar;57(1):31-7. doi: 10.1111/j.1834-7819.2011.01652.x. PMID 22369555